CLINICAL TRIAL: NCT06895655
Title: Diffusion Weighted MRI Compared to Ultrasound Elstography in the Assessment of Pancreatic Masses.
Brief Title: Mri and Ultrasound Elastography in Pancreatic Masses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousra Ahmed Osman Foley, doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRIandUSE in pancreatic masses
Record Dates: First submitted 2025-03-08; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Masses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pancreatic mass GROUP (Other)
  Interventions: Device: MRI and Ultrasound Elastography

INTERVENTIONS:
Device: MRI and Ultrasound Elastography — transcutaneous ultrasound elastography and MRI abdomen with diffusion to evaluate pancreatic mass as regard of probability of mass to be malignancy ,size of the mass ,relation to pancreatic duct and bile duct evaluation with their result will be compared to the pathologic finding.

SUMMARY:
To compare transcutaneous ultrasound elstography to Diffusion weighted MRI in differentiating between benign and malignant pancreatic masses.

DETAILED DESCRIPTION:
There are many types of pancreatic masses classified based on their nature (benign vs. malignant), type (solid vs. cystic), and histological characteristics such as pancreatic cysts, pseudocysts with pooled prevalence rate of 8%,, pancreatic ductal carcinoma (PDAC) accounts for more than 85%, neuroendocrine tumors (NET) less than 5%, and solid pseudopapillary neoplasms account for approximately 0.9%-2.7% of all exocrine pancreatic neoplasms and 5% of cystic pancreatic neoplasms. Moreover, there are some pancreatic tumorous diseases such as chronic pancreatitis and autoimmune pancreatitis .

Pancreatic cancer has a low 5-year relative survival rate of 9% .Unfortunately, the global incidence of pancreatic ductal adenocarcinoma (PDAC) is increasing by about 1% annually Presently, PDAC is the seventh leading cause of cancer-related mortality in the world, with more than 300,000 deaths reported each year.

Typically, imaging assessment is the initial process in the diagnosis of PDAC. Endoscopic ultrasonography (EUS) and/or endoscopic retrograde pancreatography may be considered as reliable tools with higher diagnostic ability. However, because of the recent trend of reducing patient burden while ensuring safety, less-invasive methods may be preferred for practical management.

Currently, the commonly used imaging examinations for pancreatic lesions include computed tomography (CT) and magnetic resonance imaging (MRI). However, despite tremendous advances in imaging, it is still challenging to accurately characterize some pancreatic lesions based on morphological imaging, such as identifying small lesions and differentiating pancreatic adenocarcinoma and mass-forming pancreatitis which represents about 5-10% of pancreatic mass cases.

Diffusion weighted imaging (DWI) is an MRI method that provides information about the microstructural characteristics of tissues by detecting the random molecular motion of water molecules and generates representative ADC values.

Diffusion-weighted imaging (DWI) provides functional information on mass tissue, like cellular density, which cannot be obtained from morphological imaging.

Previous studies showed that DWI could improve staging and prognosis evaluation of pancreatic masses and help detect small pancreatic cancers as well as differentiate pancreatic cancer from mass-forming pancreatitis.

Ultrasound elastography is a relatively new diagnostic technique for measuring tissue elasticity (hardness) by palpation.

pancreatic masses can be diagnosed using elastography as the tissue elasticities of benign and malignant tissues differ.

normally the entire pancreas has an intermediate stiffness, and the shear wave speed is about 1.4 m/sec.

There are various types of elastography devices, and each utilizes different mechanisms. In the established guideline on ultrasound elastography, the various types of elastography are classified into strain elastography, shear wave elastography, transient elastography, and acoustic radiation force impulse (ARFI) imaging.

Out of the four types of elastographies that are used in the clinical setting, strain and shear wave elastographies are mainly used in pancreatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to radiology department presented clinically with pancreatic masses and willing to participate in the study.

Exclusion Criteria:

* preoperative chemotherapy/radiotherapy cases, pancreatic stenting cases, recurrent cases after previous resection.
* patients diagnosed as acute and chronic pancreatitis
* other contraindications to MRI such as cardiac pacemaker,claustrophobia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
for shear wave elastography | 2 years
  increased shear wave speed suggesting malignancy
efficacy diffusion-weighted MRI to differentiate benigen and malignant pancreatic lesions | 2 year
  a decrease in ADC and hyperintensity signals on DWI suggesting malinant lesion
The quality evaluation for strain elastography : color pattern diagnosis is used for major color tones (blue: hard, red: soft) of tumors | 2 years
Strain ratio: high strain ratio indicate that the tumor stiffer than surrounding suggesting malignancy | 2 year

IPD SHARING:
Plan to Share IPD: Undecided